CLINICAL TRIAL: NCT04750811
Title: A Danish Audit of Small Bowel Obstruction
Acronym: DASBO
Status: Active, not recruiting | Type: Observational
Sponsor: Danish Small Bowel Obstruction Collaborative (Other)
Responsible Party: Principal Investigator, Henry Smith, Specialist Surgical Registrar, Principal Investigator, Danish Small Bowel Obstruction Collaborative
Other Study IDs: P-2021-70
Record Dates: First submitted 2021-02-03; First posted 2021-02-11 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Bowel Obstruction Small
Keywords: Small Bowel Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Small Bowel obstruction: Patients admitted with a diagnosis of small bowel obstruction at 1 of the 6 participating centres

SUMMARY:
Small bowel obstruction (SBO) is a common and potentially life-threatening acute surgical condition. A minority of patients present with a clear indication for urgent surgical intervention, either on the basis of clinical or radiological assessment (clinical signs of peritonitis/sepsis; suspicion of bowel ischaemia; closed loop obstructions; irreducible herniae etc.). However, the optimal management of the remaining patients, the majority of whom present with SBO caused by abdominal adhesions, remains a topic of international debate with practice varying in different healthcare systems.

This multicentre, prospective, observational study aims to describe the current management of patients admitted with SBO in 6 acute hospitals (Bispebjerg, Herlev, Hillerød, Hvidovre, Køge, Slagelse) on the island of Sjælland, Denmark, which accounts for a 1/3 of the total Danish population.

DETAILED DESCRIPTION:
This is a prospective, non-interventional observational study of the management and outcomes of patients admitted with SBO in Denmark.

Relevant clinicopathological demographics will be retrieved from consenting patients' medical records. An initial analysis will be performed once these patients have reached 90 days follow-up after the start of treatment. The long-term outcomes of treatment will be assessed with further analyses at 1, 3 and 5 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Radiological or clinical diagnosis of mechanical SBO
* Admitted to one of the 6 participating centres

Exclusion Criteria:

* SBO presenting within 30 days of a previous abdominal operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to participating centres on the island of Sjaelland, Denmark
Sampling Method: Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
30-day morbidity rate | 30 days
30-day mortality rate | 30 days

SECONDARY OUTCOMES:
90-day mortality rate | 90 days
To describe the proportion of patients undergoing operative versus non-operative management | From 90 days
To determine the success rate of non-operative management in patients with SBO and identify predictors of success/failure | From the start of treatment until 90-days follow-up
To determine the incidence and consequence of acute kidney injury in patients with SBO | 90 days
To determine the incidence and consequence of malnourishment in patients with SBO | 90 days

OTHER OUTCOMES:
To determine the incidence of recurrent SBO at 1-year, 3-year and 5-year follow-up. | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (6):
- Denmark (6):
  - Bispebjerg Hospital, Copenhagen, County
  - Herlev Hospital, Copenhagen
  - Hvidovre Hospital, Copenhagen
  - Hillerød Hospital, Hillerød
  - Zealand University Hospital, Køge
  - Slagelse Hospital, Slagelse

REFERENCES:
- [Derived] Mortensen MR, Alouda M, Bond Z, Burcharth J, Finne KF, Jensen TK, Lolle I, Malik T, Ngo-Stuyt L, Nielsen LBJ, Olausson M, Skovsen AP, Tolver MA, Smith HG. One-year outcomes following operative or non-operative management of adhesional small bowel obstruction. BJS Open. 2023 Sep 5;7(5):zrad103. doi: 10.1093/bjsopen/zrad103. PMID 37837353
- [Derived] Tolver MA, AErenlund MP, Azzam M, Bjerke T, Burcharth J, Dibbern CB, Jensen TK, Jordhoj JQ, Lolle I, Ngo-Stuyt L, Nielsen EO, Nielsen LBJ, Olausson M, Skovsen AP, Smith HG. Inter-hospital variation in management of patients with small bowel obstruction in Denmark. Dan Med J. 2023 Aug 16;70(9):A01230057. PMID 37622641
- [Derived] Olausson M, Aerenlund MP, Azzam M, Bjerke T, Burcharth JFH, Dibbern CB, Jensen TK, Jordhoj JQ, Lolle I, Ngo-Stuyt L, Nielsen EO, Nielsen LBJ, Skovsen AP, Tolver MA, Smith HG. Management and short-term outcomes of patients with small bowel obstruction in Denmark: a multicentre prospective cohort study. Eur J Trauma Emerg Surg. 2023 Apr;49(2):1121-1130. doi: 10.1007/s00068-022-02171-y. Epub 2022 Nov 10. PMID 36357790

DOCUMENTS (1):
  • Study Protocol (2021-02-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT04750811/Prot_001.pdf